CLINICAL TRIAL: NCT07213674
Title: A Phase 3, Open-label, Multicenter, Randomized Study of Xaluritamig Plus Abiraterone Versus Investigator's Choice in Participants With Chemotherapy-naïve Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study of Xaluritamig Plus Abiraterone Versus Investigator's Choice in Participants With Chemotherapy-naïve Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230239
Record Dates: First submitted 2025-09-18; First posted 2025-10-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate Cancer; Chemotherapy-naïve Metastatic Castration-resistant Prostate Cancer; Xaluritamig; Abiraterone; Abiraterone Acetate; Docetaxel; Cabazitaxel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Docetaxel; cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xaluritamig Plus Abiraterone (Experimental): Participants will be randomized to receive xaluritamig in combination with abiraterone acetate.
  Interventions: Drug: Xaluritamig; Drug: Abiraterone acetate
- Investigator's Choice (Active Comparator): Participants will receive investigator's choice of:
  * Abiraterone acetate orally, once daily or
  * Docetaxel IV Q3W or
  * Cabazitaxel IV Q3W.
  Interventions: Drug: Abiraterone acetate; Drug: Docetaxel; Drug: Cabazitaxel

INTERVENTIONS:
Drug: Xaluritamig — Xaluritamig will be administered IV.
  Other Names: AMG 509
  Arms: Xaluritamig Plus Abiraterone
Drug: Abiraterone acetate — Abiraterone acetate will be administered orally.
Drug: Docetaxel — Docetaxel will be administered IV.
  Arms: Investigator's Choice
Drug: Cabazitaxel — Cabazitaxel will be administered IV.
  Arms: Investigator's Choice

SUMMARY:
The primary objective of this study is to compare overall survival (OS) in participants receiving xaluritamig plus abiraterone against investigator's choice (docetaxel, cabazitaxel, or abiraterone).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent before initiation of any study-specific activities/procedures.
* Age ≥ 18 years (or ≥ legal age within the country if it is older than 18 years) at the time of signing the informed consent.
* Participant must have histological, pathological, and/or cytological confirmation of adenocarcinoma of the prostate. Mixed histologies (eg, adenocarcinoma with neuroendocrine component) are not permitted.
* Metastatic castration-resistant prostate cancer (mCRPC) with ≥ 1 metastatic lesion that is present on baseline computed tomography (CT), magnetic resonance imaging (MRI), or bone scan imaging obtained within 28 days before enrollment.
* Evidence of progressive disease (PD), defined as 1 or more PCWG3-modified RECIST 1.1 criteria:

  * Serum PSA progression is defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week prior. The minimum start value is 2.0 ng/mL.
  * Soft-tissue progression defined as an increase ≥ 20% in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since treatment started or the appearance of 1 or more new lesions or unequivocal progression of existing non-target lesions.
  * Progression of bone disease defined by the appearance of at least 2 new bone lesions(s) by bone scan (as per the 2+2 PCWG3-modified RECIST 1.1 criteria).
* Participants must have had prior orchiectomy and/or ongoing androgen-deprivation therapy (ADT) and a castrate level of serum testosterone (< 50 ng/dL or < 1.7 nmol/L).
* Prior disease progression on 1, and only 1, androgen receptor pathway inhibitor (ARPI) (either enzalutamide, apalutamide, or darolutamide) is required.
* Participants intended to receive cabazitaxel must have previously received ≤ 6 cycles of docetaxel in the metastatic hormone-sensitive prostate cancer (mHSPC) setting.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Adequate organ function.

Exclusion Criteria:

Disease Related:

* Participants with a history of central nervous system (CNS) metastases.
* Unresolved toxicities from prior antitumor therapy not having resolved to CTCAE version 5.0 grade 1 or baseline, with the exception of alopecia or toxicities that are stable and well-controlled AND there is an agreement to allow inclusion by both the investigator and the sponsor.

Prior/Concomitant Therapy:

* Prior six transmembrane epithelial antigen of the prostate 1 (STEAP1)-targeted therapy.
* Prior disease progression on or intolerance to abiraterone.
* Prior treatment with any chemotherapy regimen in the mCRPC setting and/or > 6 cycles of docetaxel treatment in the mHSPC setting.
* Any anticancer therapy, immunotherapy, or investigational agent within 4 weeks before first dose of study treatment with the following exceptions:

  * Androgen receptor pathway inhibitors (ARPIs; enzalutamide, darolutamide, apalutamide): minimum washout of 2 weeks prior to the first dose of study treatment.
  * Androgen suppression therapy (eg, luteinizing hormone-releasing hormone/gonadotrophin releasing hormone [LHRH/GnRH] analogue [agonist/antagonist]) is permitted.
* Prior radioligand therapy (RLT) within 8 weeks of first dose of study treatment.
* Prior radionuclide therapy (radium-223) within 2 months of first dose of study treatment.
* Prior palliative radiotherapy within 2 weeks before first dose of study treatment. Participants must have recovered from all radiation-related toxicities.
* Concurrent cytotoxic chemotherapy, ARPI, immunotherapy, RLT, poly adenosine diphosphate ribose polymerase (PARP) inhibitor, biological therapy, investigational therapy.
* Treatment with live and live-attenuated vaccines within 4 weeks before the first dose of study treatment.
* Prior CD3-directed therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2030-01-07 (Estimated); Study Completion 2032-08-30 (Estimated)

PRIMARY OUTCOMES:
OS | Up to approximately 51 months

SECONDARY OUTCOMES:
Radiographic Progression-free Survival (rPFS) Per Prostate Cancer Working Group 3 (PCWG3)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), Per Investigator Assessment | Up to approximately 51 months
Objective Response per Modified RECIST 1.1, Per Investigator Assessment | Up to approximately 51 months
Duration of Response (DOR) Per Modified RECIST 1.1, Per Investigator Assessment | Up to approximately 51 months
Disease Control Per Modified RECIST 1.1, Per Investigator Assessment | Up to approximately 51 months
Progression-free Survival (PFS) 2, Per Investigator Assessment | Up to approximately 51 months
Time to Response (TTR), Per Modified RECIST 1.1, Per Investigator Assessment | Up to approximately 51 months
Time to First Subsequent Therapy | Up to approximately 51 months
Time to Symptomatic Skeletal Events (SSE) | Up to approximately 51 months
Number of Participants With Treatment-emergent Adverse events, Treatment-emergent Serious Adverse Events, and Fatal Adverse Events | Up to approximately 51 months
Change From Baseline Over Time at Each Assessment in Brief Pain Inventory - Short Form (BPI-SF) Pain Intensity Scale | Up to approximately 51 months
Change From Baseline Over Time at Each Assessment in BPI-SF Worst Pain Score | Up to approximately 51 months
Change From Baseline Over Time at Each Assessment in BPI-SF Pain Interference Scale | Up to approximately 51 months
Change From Baseline Over Time at Each Assessment in Functional Assessment of Cancer Therapy - Prostate (FACT-P) Total Score and Subscale Scores | Up to approximately 51 months
Change From Baseline Over Time at Each Assessment in European Quality of Life (EuroQol) 5 Domain 5 Level Scale (EQ-5D-5L) Utility Score | Up to approximately 51 months
Change From Baseline Over Time at Each Assessment in the EQ-5D-5L Visual Analogue Scale (VAS) | Up to approximately 51 months
Time to Worsening as Measured by BPI-SF Worst Pain Score | Up to approximately 51 months
Time to Worsening as Measured by BPI-SF Pain Intensity Scale | Up to approximately 51 months
Time to Worsening as Measured by BPI-SF Pain Interference Scale | Up to approximately 51 months
Time to Worsening as Measured by FACT-P Total Score | Up to approximately 51 months
Time to Improvement as Measured by BPI-SF Worst Pain Score in Participants with Moderate/Severe Pain at Baseline | Up to approximately 51 months
Time to Improvement After Worsening as Measured by BPI-SF Pain Intensity Scale Score | Up to approximately 51 months
Time to Improvement After Worsening as Measured by BPI-SF Pain Interference Scale Score | Up to approximately 51 months
Summary Scores Over Time at Each Assessment as Measured by Selected Questions on Symptomatic Adverse Events from the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Item Library | Up to approximately 51 months
Summary Scores Over Time at Each Assessment as Measured by the GP5 Question on Overall Bother of Side Effects from the FACT-P Questionnaire | Up to approximately 51 months
Prostate-specific Antigen (PSA) 50 and PSA 90 Responses | Up to approximately 51 months
Time to PSA 50 and PSA 90 Response | Up to approximately 51 months
Duration of PSA 50 and PSA 90 Response | Up to approximately 51 months
Time to PSA Progression | Up to approximately 51 months
Maximum Serum Concentration (Cmax) of Xaluritamig | Up to approximately 51 months
Time to Maximum Concentration (Tmax) of Xaluritamig | Up to approximately 51 months
Minimum Serum Concentration (Cmin) of Xaluritamig | Up to approximately 51 months
Area Under the Concentration-time Curve (AUC) Over the Dosing Interval of Xaluritamig | Up to approximately 51 months
Accumulation Ratio of the AUC Over the Dosing Interval for Xaluritamig | Up to approximately 51 months
Half-life (t1/2) of Xaluritamig | Up to approximately 51 months
Abiraterone Serum Concentrations | Up to approximately 51 months
Number of Participants with Formation of Anti-xaluritamig Antibodies | Up to approximately 51 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (79):
- United States (10):
  - City of Hope National Medical Center, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Duarte, California
  - Providence Saint Jude Medical Center, Fullerton, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - University of Illinois Chicago, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Hightower Clinical, Oklahoma City, Oklahoma
  - United States Oncology Regulatory Affairs Corporate Office, Nashville, Tennessee
  - US Oncology Research Investigational Products Center, Tyler, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
- Australia (5):
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Icon Cancer Care Wesley, Herston, Queensland
  - Tasman Oncology Research, Southport, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Austin Hospital, East Melbourne, Victoria
- Austria (3):
  - Universitaetsklinikum Sankt Poelten, Sankt Pölten
  - Krankenhaus der Barmherzigen Brueder Wien, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Belgium (2):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
- France (3):
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Saint Andre, Bordeaux
  - Centre Leon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
- Germany (9):
  - Charite - Universitaetsmedizin Berlin, Campus Mitte, Berlin
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Jena, Jena
  - Universitaetsklinikum Schleswig-Holstein - Kiel, Kiel
  - Universitaetsklinikum Ulm, Ulm
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (5):
  - Alexandra Hospital, Athens
  - University Hospital of Heraklion, Heraklion - Crete
  - General Oncological Hospital of Kifisia Oi Agioi Anargyroi, Kifissia, Athens
  - Athens Medical Center S.A - Iatriko Amarousiou, Marousi
  - European Interbalkan Medical Center, Thessaloniki
- Italy (5):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - Ospedale Santa Chiara Azienda Provinciale per i Servizi Sanitari Provincia Autonoma di Trento, Trento
- Japan (13):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kobe University Hospital, Kobe, Hyōgo
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Osaka International Cancer Institute, Osaka, Osaka
  - The University of Osaka Hospital, Suita-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Dokkyo Medical University Saitama Medical Center, Koshigaya-shi, Saitama
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - The Cancer institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Portugal (3):
  - Hospital da Luz, SA, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saude de Sao Joao, EPE - Hospital de Sao Joao, Porto
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (7):
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (4):
  - Inselspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Sankt Gallen, Sankt Gallen
  - Hirslanden Zurich, Zurich
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
- United Kingdom (2):
  - Sarah Cannon Research Institute UK, London
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com